CLINICAL TRIAL: NCT05799573
Title: CT-scan Sizing Perceval Sutureless Valve
Brief Title: CT Scan Sizing for Perceval Sutureless Valve
Acronym: PERCEVAL
Status: Recruiting | Type: Observational
Sponsor: Maria Cecilia Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PERCEVAL
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Aortic Valve Regurgitation
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Perceval sutureless aortic bioprosthesis is a bovine pericardium valve mounted in a nitinol stent that can be compressed and positioned in a valve delivery system. Similarly, to transcatheter aortic valve implantation (TAVI) devices, the anchoring and good sealing of the Perceval bioprosthesis relies on oversizing by design of the nitinol stent compared with the native aortic annulus. With the advent of TAVI, cardiac computed tomography (CT) has become the gold standard technique for measuring the aortic annulus in patients undergoing transcatheter procedures, and the CT-derived axial image of the aortic virtual basal ring (VBR) is considered as the reference for sizing by most of the manufacturers of transcatheter valves .

Interestingly, the VBR lies exactly on the plane passing through the nadir of the 3 aortic cusps, that is where, according to the instructions for use, a correctly positioned Perceval valve should be deployed. VBR could then provide a good estimate of the annular dimension for the Perceval pre-operative sizing.

DETAILED DESCRIPTION:
Recent evidence in TAVI patients suggests that significant underexpansion or distortion of valved stents may be associated with altered leaflet function, leading to increased transprosthetic gradients and possibly predisposing to other negative outcomes such as valve thrombosis, low platelet counts, thromboembolic events, and early degeneration . Moreover, there is evidence that excessive oversizing of the Perceval valve is detrimental.

The present study is aimed to investigate the relationship between the CT-derived measure of the annulus dimension and early hemodynamic and clinical outcomes in patients undergoing sutureless aortic valve replacement (AVR) with the Perceval sutureless aortic valve and define the Perceval sizing chart based on preoperative CT-scan measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects > 18 years;
2. Subjects willing to sign and date an informed consent for treatment of personal data;
3. Subjects willing and able to comply with the follow up schedule of the protocol;
4. Subjects with indication for aortic valve replacement on a tricuspid aortic valve;
5. Subjects with possibly associated need for coronary revascularization.
6. Subjects with Ejection Fraction ≥ 40%

Exclusion Criteria:

1. Male and female subjects ≤ 18 years;
2. Subjects with bicuspid aortic valve
3. Subjects with associated mitral valvulopathy or ascending aorta aneurysm
4. Subjects with pure aortic insufficiency
5. Subjects with Ejection Fraction < 40%
6. Subjects with acute myocardial infarction < 30 gg
7. Subjects with serum creatinine > 2 mg/Dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indication for aortic valve replacement with a Perceval valve
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the proper Perceval valve size assessed by the early postoperative outcomes at discharge | 12 months
  The primary endpoint is to evaluate the proper Perceval valve size assessed by the early postoperative outcomes at discharge in terms of:
  * Mean and peak pressure gradients
  * Prosthetic regurgitation
  * migration/dislodgement
  * need for permanent pacemaker implant

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Mikus, MD, Principal Investigator — Maria Cecilia Hospital
Locations (1):
- Maria Cecilia Hospital, Cotignola, Ravenna, Italy

IPD SHARING:
Plan to Share IPD: No
All information related to the participation of a subject in this study will be treated with the utmost confidentiality, in accordance with good clinical practice (Decree of the Ministry of Health of 15 July 1997, and subsequent amendments and additions) and regulations on the protection of personal data: Information and Consent pursuant to Legislative Decree no. 196 of 30/06/2003 and the European General Data Protection Regulation (GDPR - General Data Protection Regulation), which came into force on 25 May 2018.
  All patient names will be kept confidential. Patients will be identified throughout documentation and evaluation by the number allotted to them by the study. The patients will be assured that all findings will be stored on computer and handled in the strictest confidence. The Investigator agrees to maintain the confidentiality of the study protocol.